CLINICAL TRIAL: NCT06322836
Title: Electra-1; Elective Cardioversion of Atrial Fibrillation at Home by Advanced Practice Providers; A Feasibility Study in Dutch Emergency Medical Service
Brief Title: A Feasibility Study for Elective Cardioversion of Atrial Fibrillation at Home
Acronym: Electra-1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RAV Brabant MWN (Other)
Collaborators: Jeroen Bosch Ziekenhuis (Other)
Responsible Party: Principal Investigator, Risco van Vliet, Principal Investigator, RAV Brabant MWN
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Protocol ID ABR number 83536
Record Dates: First submitted 2024-02-27; First posted 2024-03-21 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Emergency Medical Services; Electric Countershock
Keywords: atrial fibrilation; DC-ECV

STUDY DESIGN:
Intervention Model Description: a pilot, non-controlled, non-randomised, single centre study. The Electra-1 pilot study is a prospective intervention feasibility study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- intervention arm (Other): there is only one intervention arm
  Interventions: Procedure: Duble current electro cardioversion

INTERVENTIONS:
Procedure: Duble current electro cardioversion — Instead of the regular clinical treatment, in this study direct-current electrical cardioversion (DC-ECV) will be performed at the patient's home and will be carried out by well-trained and certified advanced practice providers (APP) on site, i.e. nurse practitioner or physician assistant, supported by an EMS ambulance team containing an ambulance nurse and ambulance driver, both trained advanced life-support (ALS) professionals.

SUMMARY:
The goal of this pilot, non-controlled, non-randomised, single centre, prospective intervention feasibility study is to assess the feasibility of a home DC-ECV in the treatment of recurrent symptomatic AF performed by APP in 25 patients.

The main question[s] it aims to answer are:

Primary objective:

In this prospective intervention feasibility study, in 25 patients the primary endpoint is completion of cardioversion to sinus rhythm. (% of study patients with a recurrence of AF in whom a home cardioversion is performed, i.e. to whom at least one DC shock was administered while the patient was under sedation).

Feasibility endpoints are ; (a) evaluation of enrolment of participants, (b) evaluation and refinement of data and outcome collection procedures, (c) evaluation of logistics, (d) evaluation of the appropriateness of the intervention and research procedures to manage and implement the intervention, and (e) preliminary evaluation of participant responses to the intervention.

Secondary objectives:

Safety endpoint:

Complications immediately during and one hour after cardioversion (e.g. arrhythmias, changes in the electrocardiogram, hypotension related to sedation and/or vasodilation or skin irritation).

A composite of major adverse cardiovascular and cerebrovascular events (MACCE) occurring within 24 hours MACCE occurring during 6 weeks follow-up; any hospitalisation and all-cause mortality during 6 weeks follow-up; number (%) of patients in sinus rhythm at 1 hour in the post-shock observation period; idem at the end of 6 weeks follow-up; inventory of all interventions in the study related to cost-of-care.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent.
2. Age 18 -75 year subjects, able to understand the provided information and sign an informed consent.
3. Need for direct current electrical cardioversion (DC-ECV) for correction of recurrent symptomatic AF (according to the guidelines of the American College of Cardiology/American Heart Association/European Society of Cardiology (ACC/AHA/ESC)).
4. Weight more than 50 kilograms.
5. Successful hospital DC-ECV for a previous episode of AF performed under propofol sedation.
6. Target range of international normalized ratio (INR) above 2.0, when on vitamin K antagonists, or use of novel oral anticoagulant, stable for 3 weeks.
7. ASA 2.
8. BMI < 35 kg/m2.
9. Fasting status: at least 6 hours for food, and 2 hours for fluids.

Exclusion Criteria:

* 1. Patients over 75 years old and younger than 18 years. 2. Patients wearing pacemaker or implantable cardioverter-defibrillator. 3. Patients with (cardiovascular): sick sinus syndrome, ventricular pre-excitation, Brugada syndrome or bundle branch block.

severe ischemic or valvular heart disease. known second or third degree atrioventricular block normal sinus rhythm. heart failure NYHA III or IV, known LVEF < 35%, or cor pulmonale. transient and reversible cause of AF, e.g. in setting of fever and hyperthyroidism.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2024-02-07 (Actual); Primary Completion 2024-08-29 (Actual); Study Completion 2025-02-10 (Actual)

PRIMARY OUTCOMES:
completion of cardioversion to sinus rhythm | within 60 minutes after cardioversion
  % of study patients with a recurrence of AF in whom a home cardioversion is performed, i.e. to whom at least one DC shock was administered while the patient was under sedation

SECONDARY OUTCOMES:
Incidence of treatment-emergent adverse events (Safety endpoint a) | up to 1 hour after treatment
  Complications immediately during and one hour after cardioversion (e.g. arrhythmias, changes in the electrocardiogram, hypotension related to sedation and/or vasodilation or skin irritation).
Incidence of treatment-emergent adverse events (Safety endpoint b) | during 6 weeks follow-up
  A composite of major adverse cardiovascular and cerebrovascular events (MACCE) during 6 weeks follow-up; any hospitalisation and all-cause mortality during 6 weeks follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Risco V Vliet, MSc, Principal Investigator — https://www.ravbrabantmwn.nl
Locations (1):
- RAV Brabant MWN, 's-Hertogenbosch, North Brabant, Netherlands

REFERENCES:
- [Derived] van Vliet R, van Eck M, Wieringa WG, Moors XRJ, van 't Hof AWJ. Elective cardioversion of atrial fibrillation at home by advanced practice providers: a feasibility study in the Dutch emergency medical service-design and pilot results. Eur J Cardiovasc Nurs. 2025 Dec 29;24(8):1324-1330. doi: 10.1093/eurjcn/zvaf140. PMID 40674510